Clinical research protocol

Project name: The value of critical care ultrasound and

noninvasive cardiac output monitoring in guiding fluid resuscitation

for septic shock in the emergency department

leading unit:Guangzhou Panyu Central Hospital, Guangzhou,

Guangdong, China

project leader:Xiaowei Mai

Department: Emergency Department

Research period: July 2025 to July 2025

Version No.: V 1.0

Version Date: May 22, 2023

| object name | The value of critical care ultrasound and non-invasive cardiac output |
|---|---|
| | monitoring in fluid resuscitation for emergency department patients with |
| | septic shock. |
| goal of study | This study explores the value of critical care ultrasound and |
| | non-invasive cardiac output monitoring in fluid resuscitation for emergency |
| | department patients with septic shock, providing evidence for optimizing |
| | hemodynamic management of septic shock, improving patient prognosis, and |
| | guiding clinical selection of appropriate monitoring modalities. |
| research design | Subjects were recruited from patients with septic shock admitted to the |
| | Emergency Department of Guangzhou Panyu District Central Hospital |
| | between July 2023 to luly 2025. Demographic data of patients, including |
| | gender, age, and underlying diseases, were collected, along with mean |
| | arterial pressure, baseline lactate levels, and vital signs at enrollment. |
| | Records were made of the total fluid volume administered within the first 6 |
| | hours after patients were randomized into groups, the achievement of |
| | resuscitation targets, blood lactate levels, blood pressure, and the incidence of |
| | complications such as pulmonary edema and renal injury. Additionally, the |
| | use of vasoactive agents (e.g., dopamine, epinephrine/norepinephrine), |
| | mechanical ventilation support, and antibiotics was documented. Patients |
| | were followed up to record the duration of emergency department stay, total |
| | hospital stay, 28-day mortality, and adverse events occurring during the study |
| | period (e.g., severe arrhythmias, anaphylactic shock). |
| Total number of | |
| | 60 cases (30 cases in each group) |
| cases studied | |

#### Inclusion criteria:

(1) diagnosis of septic shock in accordance with the Surviving Sepsis
 Campaign International; (2) receipt of initial fluid resuscitation in the
 emergency department with a hospital stay of at least 6 hours; (3) age ≥ 18
 years; (4) provision of informed consent.

## case selection

## excluded criteria:

(1) contraindications to rapid fluid administration (e.g., end-stage renal disease, end-stage heart failure, acute pulmonary edema); (2) inability to comply with treatment, such as patients with severe trauma, burns, cancer undergoing chemotherapy, pregnant or lactating women, and those with mental illness; (3) withdrawal from treatment or transfer to another facility within 24 hours of admission.

## Treatment plan

Both groups were managed according to the 2021 Surviving Sepsis Campaign (SSC) International Guidelines for septic shock resuscitation, including: (1) early antimicrobial therapy, (2) vasopressor support (with norepinephrine as first-line), and (3) organ function support. The key difference between groups lay in the fluid resuscitation monitoring approach (critical care ultrasound vs. noninvasive cardiac output monitoring)

# efficacy evaluation

The main efficacy indicators: emergency department length of stay, total hospital stay.

Secondary efficacy indicators: regarding total fluid volume within the first 6 hours of resuscitation, early resuscitation efficacy (time to achieve mean arterial pressure  $\geq$ 65 mmHg, lactate reduction  $\geq$ 20% from baseline, or lactate clearance  $\geq$  10%), complication rates (including pulmonary edema, renal injury, and acute respiratory distress syndrome).

Safety evaluation index: 28-day mortality.

#### statistical method

This study adopted a prospective randomized controlled design, and the sample size was estimated using PASS 15.0 software. Based on the difference in 6-hour fluid resuscitation volume between the two groups in the pilot study (mean difference 1261 mL, standard deviation 3155 mL), α=0.05 (bilateral) was set  $\beta$ =0.2, Calculated to require 27 cases per group, considering a 20% dropout rate, 60 cases were ultimately included. Use SPSS 26.0 to generate block random sequences (block size 4), and allocate concepts through sealed envelopes. The normality of the measurement data was confirmed by Shapiro Wilk test, and those that conform to the normal distribution were expressed as mean ± standard deviation. Independent sample t-test was used for inter group comparison; non normally distributed individuals are represented by the median (interquartile range) and Mann Whitney U test is used. The categorical data is presented in terms of the number of cases (%), and the comparison between groups is conducted using the chi square test or Fishers exact test (when the theoretical frequency is less than 5). The main outcome (28 day mortality rate) was plotted using Kaplan Meier survival curve, and inter group differences were analyzed using log rank test, and HR (95% CI) was calculated. Secondary outcomes (such as fluid dosage, MAP, etc.) report mean difference (MD) or relative risk (RR) and their 95% confidence intervals. All tests are bilateral, and P<0.05 is considered statistically significant. Perform Bonferroni correction on secondary outcomes ( $\alpha$ =0.05/6  $\approx$  0.008). Multivariate Cox regression was used to adjust for confounding factors such as age and baseline lactate, and sensitivity analysis included protocol set (PP) and intention to treat (ITT) analyses. The statistical software used is R 4.3.1 (R Foundation) and SPSS 26.0 (IBM).

| Research period | July 2023 to luly 2025 |
|-----------------|------------------------|
|-----------------|------------------------|

#### (1)Research background

Septic shock represents the severe phase of infection-induced systemic inflammatory response syndrome (SIRS), characterized by a complex pathophysiological mechanism. It is primarily manifested as vasodilation, capillary leakage, and myocardial depression triggered by SIRS, with persistent hypotension, tissue hypoperfusion, and multiple organ dysfunction resulting from insufficient effective circulating blood volume as the main clinical features. With a mortality rate exceeding 40%, it ranks among the common critical illnesses in the emergency department. International guidelines for the management of septic shock highlight that early goal-directed fluid resuscitation is the cornerstone of septic shock treatment. It aims to alleviate the systemic damage caused by shock by rapidly restoring effective circulating blood volume and increasing tissue oxygen delivery, thereby improving prognosis and enhancing quality of life. Consequently, fluid resuscitation holds an irreplaceable role in the management of septic shock, and the first 6 hours after shock recognition, in particular, is designated as the "golden resuscitation period". However, both excessive and insufficient fluid resuscitation may exacerbate the condition and elevate the risk of complications such as pulmonary edema, acute respiratory distress syndrome (ARDS), and acute kidney injury (AKI). Thus, how to rapidly and accurately assess a patients volume status and cardiac function in the emergency department, formulate individualized fluid resuscitation strategies, achieve precise volume management, and avoid over-resuscitation or under-resuscitation has become an urgent clinical challenge.

Traditional fluid resuscitation strategies rely predominantly on static parameters such as central venous pressure (CVP), mean arterial pressure (MAP), and urine output for guidance. However, these indices have inherent limitations in assessing volume responsiveness and predicting fluid resuscitation efficacy, failing to accurately and dynamically reflect a patients volume status or cardiac preload responsiveness. In recent years, with advances in hemodynamic monitoring technologies, dynamic evaluation of volume responsiveness has emerged as a key strategy for optimizing fluid resuscitation and improving patient outcomes.

Critical care ultrasound, for instance, enables rapid bedside assessment of cardiopulmonary function by real-time visualization of indices including inferior vena cava variability, ventricular wall motion, volume responsiveness, and lung water content, thereby providing visual evidence to guide early fluid resuscitation. Non-invasive cardiac output monitoring, conversely, dynamically tracks circulatory function through quantification of parameters such as cardiac output and stroke volume variability, offering objective data to evaluate resuscitation efficacy. Accordingly, critical care ultrasound and non-invasive cardiac output monitoring have increasingly become valuable clinical adjuncts in guiding fluid resuscitation for patients with septic shock in the emergency department.

## (2) research objective

- 1. Main Objective: This study explores the value of critical care ultrasound and non-invasive cardiac output monitoring in fluid resuscitation for emergency department patients with septic shock, providing evidence for optimizing hemodynamic management of septic shock, improving patient prognosis, and guiding clinical selection of appropriate monitoring modalities.
- 2.Secondary purpose: This study aims to explore the value of critical care ultrasound and non-invasive cardiac output monitoring in fluid resuscitation for emergency department patients with septic shock, to inform optimized hemodynamic management, improve prognosis, and guide clinical selection of monitoring modalities.

#### (3) Research Design Types, Principles, and Test Procedures

### 1. Research Design

Subjects were recruited from patients with septic shock admitted to the Emergency Department of Guangzhou Panyu District Central Hospital between July 2023 to luly 2025. Demographic data ofpatients, including gender, age, and underlying diseases, were collected, along with mean arterial pressure, baseline lactate levels, and vital signs at enrollment. Records were made of the total fluid volume administered within the first 6 hours after patients were randomized into groups, the achievement of resuscitation targets,

blood lactate levels, blood pressure, and the incidence of complications such as pulmonary edema and renal injury. Additionally, the use of vasoactive agents (e.g., dopamine, epinephrine/norepinephrine), mechanical ventilation support, and antibiotics was documented. Patients were followed up to record the duration of emergency department stay, total hospital stay, 28-day mortality, and adverse events occurring during the study period (e.g., severe arrhythmias, anaphylactic shock).

After patients met the inclusion criteria and signed the informed consent form, random numbers were generated using SPSS 26.0 statistical software to randomly assign 73 participants to the critical care ultrasound group and the non-invasive cardiac output group. The generated random allocation table was prepared in duplicate, which were sealed and stored by the statistician and research coordinator respectively to prevent premature disclosure of group allocation information.

In the critical care ultrasound group, patients underwent immediate bedside assessment using a Philips EPIQ 5 color Doppler ultrasound system equipped with both phased-array (1.5-4.0 MHz) and convex-array (2.0-5.0 MHz) transducers. The initial ultrasound evaluation was completed within 10 minutes of enrollment and included comprehensive hemodynamic monitoring: inferior vena cava diameter (IVC) and collapsibility index (IVC-CI) for volume status assessment, left ventricular ejection fraction (LVEF) and end-diastolic volume (LVEDV) for cardiac function evaluation, ventricular wall motion analysis, along with pulmonary B-line quantification to assess pulmonary edema. This protocol ensured real-time, comprehensive evaluation of both cardiac function and fluid status to guide resuscitation. Ultrasound reassessment was performed every 1-2 hours to dynamically adjust both the volume and rate of fluid administration until predefined resuscitation targets were achieved.

In the noninvasive cardiac output monitoring group, continuous hemodynamic assessment was performed using the NICOM system based on thoracic bioreactance technology. Following the manufacturers standard operating procedures, four electrode pads were placed at bilateral subclavicular areas and the left subcostal region. Monitoring commenced immediately after

enrollment, with baseline parameters recorded after signal stabilization (≤5 minutes), including cardiac output (CO), stroke volume (SV), stroke volume variation (SVV), and systemic vascular resistance (SVR). The system automatically updated these parameters every 30 seconds and displayed them in real-time on the monitor screen. Fluid resuscitation was dynamically adjusted according to these continuous measurements until achieving the predefined therapeutic targets.

#### (4) case selection

- 1. Inclusion criteria:
- (1) diagnosis of septic shock in accordance with the Surviving Sepsis Campaign International; (2) receipt of initial fluid resuscitation in the emergency department with a hospital stay of at least 6 hours; (3) age  $\geq$  18 years; (4) provision of informed consent.

#### 2. excluded criteria:

(1) contraindications to rapid fluid administration (e.g., end-stage renal disease, end-stage heart failure, acute pulmonary edema); (2) inability to comply with treatment, such as patients with severe trauma, burns, cancer undergoing chemotherapy, pregnant or lactating women, and those with mental illness; (3) withdrawal from treatment or transfer to another facility within 24 hours of admission.

#### 3. Elimination criteria

Subjects who have been enrolled in the study but meet one ofthe following criteria should be excluded:

- ( 1) After inclusion, those who did not meet the inclusion criteria or met the exclusion criteria were found.
  - (2) Those who have not used test drugs / interventions.
  - 4. Standard for suspension of research
- (1) If the following conditions occur during the experiment: cardiac arrest, intestinal perforation, intracranial and other serious complications; (2) the need for rescue is not suitable for experimental related operators; (3) The competent physician believes that the clinical condition is not suitable for continuing the experiment; (4) If the clinical symptoms

and other auxiliary examinations are inconsistent with the relevant non-invasive examination results; (5) Someone did not agree to continue the experiment during the experiment.

#### 5 . Drop-out / exit criteria

Expulsion / withdrawal criteria: ( 1 ) the competent physician believes that the clinical condition is not suitable for the continuation of the experiment; ( 2 ) If the clinical symptoms and other auxiliary examinations are inconsistent with the relevant non-invasive examination results; ( 3 ) Someone did not agree to continue the experiment during the experiment.

## (5)research method

Subjects were recruited from patients with septic shock admitted to the Emergency Department of Guangzhou Panyu District Central Hospital between December 2022 and January 2026. Demographic data of patients, including gender, age, and underlying diseases, were collected, along with mean arterial pressure, baseline lactate levels, and vital signs at enrollment. Records were made of the total fluid volume administered within the first 6 hours after patients were randomized into groups, the achievement of resuscitation targets, blood lactate levels, blood pressure, and the incidence of complications such as pulmonary edema and renal injury. Additionally, the use of vasoactive agents (e.g., dopamine, epinephrine/norepinephrine), mechanical ventilation support, and antibiotics was documented. Patients were followed up to record the duration of Emergency Department stay, total hospital stay, 28-day mortality, and adverse events occurring during the study period (e.g., severe arrhythmias, anaphylactic shock).

## (6) Observation items and detection time points

- Demographic data of patients, including gender, age, and underlying diseases, were collected, along with mean arterial pressure, baseline lactate levels, and vital signs at enrollment.
- 2. Records were made ofthe total fluid volume administered within the first 6 hours after patients were randomized into groups, the achievement of resuscitation targets, blood

lactate levels, blood pressure, and the incidence of complications such as pulmonary edema and renal injury.

- 3. Document the use of vasoactive agents (e.g., dopamine, epinephrine/norepinephrine), mechanical ventilation support, and antibiotics.
- 4. Record the duration of Emergency Department stay, total hospital stay, 28-day mortality, and adverse events occurring during the study period (e.g., severe arrhythmias, anaphylactic shock).

# (7) standards for efficacy appraisal

The primary outcome was 28-day mortality

Secondary outcomes included the efficacy of initial resuscitation, duration of hospital stay, incidence of complications, and other relevant parameters.

## (8) Observation of adverse events

Observation of adverse events: Clinicians should evaluate the fluid resuscitation of children at any time during the experiment. If the clinical symptoms and other auxiliary examinations ( such as heart rate, liver size, mental state, X-ray, blood gas analysis, etc. ) If they are inconsistent with the relevant non-invasive examinations, the experiment should be terminated immediately and the superior physician should be found in time to assist.

# (9)Data security monitoring

Clinical research will develop a corresponding data security monitoring plan based on the size ofthe risk. All adverse events were recorded in detail, properly handled and tracked until they were properly resolved or stable. Serious adverse events and unexpected events were reported to the ethics committee, competent authorities, sponsors and drug supervision and management departments in a timely manner according to the regulations. The main researchers regularly conduct a cumulative review of all adverse events, and if necessary, convene a meeting of researchers to assess the risks and benefits ofthe study; research that is greater than the minimum risk will arrange independent data monitors to monitor the research data, and high-risk research will establish an independent data security supervisory

committee to monitor the accumulated security data and effectiveness data to make recommendations on whether the research will continue.

# (10)Statistical processing

This study adopted a prospective randomized controlled design, and the sample size was estimated using PASS 15.0 software. Based on the difference in 6-hour fluid resuscitation volume between the two groups in the pilot study (mean difference 1261 mL, standard deviation 3155 mL),  $\alpha$ =0.05 (bilateral) was set  $\beta$ =0.2, Calculated to require 27 cases per group, considering a 20% dropout rate, 60 cases were ultimately included. Use SPSS 26.0 to generate block random sequences (block size 4), and allocate concepts through sealed envelopes. The normality of the measurement data was confirmed by Shapiro Wilk test, and those that conform to the normal distribution were expressed as mean ± standard deviation. Independent sample t-test was used for inter group comparison; non normally distributed individuals are represented by the median (interquartile range) and Mann Whitney U test is used. The categorical data is presented in terms of the number of cases (%), and the comparison between groups is conducted using the chi square test or Fishers exact test (when the theoretical frequency is less than 5). The main outcome (28 day mortality rate) was plotted using Kaplan Meier survival curve, and inter group differences were analyzed using log rank test, and HR (95% CI) was calculated. Secondary outcomes (such as fluid dosage, MAP, etc.) report mean difference (MD) or relative risk (RR) and their 95% confidence intervals. All tests are bilateral, and P<0.05 is considered statistically significant. Perform Bonferroni correction on secondary outcomes ( $\alpha$ =0.05/6  $\approx$  0.008). Multivariate Cox regression was used to adjust for confounding factors such as age and baseline lactate, and sensitivity analysis included protocol set (PP) and intention to treat (ITT) analyses. The statistical software used is R 4.3.1 (R Foundation) and SPSS 26.0 (IBM).

## (11) Ethics in clinical research

Clinical research will follow the World Medical Congress Helsinki Declaration and other relevant provisions. Before the study began, the clinical study was carried out after the

ethics committee approved the test plan. Before each subject is selected for this study, the researcher has the responsibility to fully and comprehensively introduce the purpose, procedure and possible risks ofthis study to the subjects or their agents, and to sign a written informed consent form. The subjects should be informed that they have the right to withdraw from the study at any time. Informed consent should be retained as a clinical research document for review. The personal privacy and data confidentiality of the subjects will be protected during the study.

#### (12)Research progress

From June 2023 to june 2023: Preparation stage for the experiment: ① Prepare relevant instruments and equipment, as well as equipment maintenance, testing, and parameter calibration; ② Recruitment and training of staff, clear division of labor and job responsibilities, and familiarity with the experimental process; ③ Complete the pre experiment.

From july 2023 to july 2025: Recruit research subjects and conduct clinical trials. ①
Recruit research subjects and implement interventions in groups according to the randomization plan; ② Record the relevant data of the experiment and follow up on the prognosis for 28 days.

From July 2025 to December 2025: Organize research data and conduct statistical analysis; Writing and submitting research papers. Summarize research results and write a project summary report.

#### (13) Reference

- [1] Fleischmann C, Scherag A, Adhikari NK, et al. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016; 193(3):259-272. doi:10.1164/rccm.201504-0781OC.
- [2] Vincent JL, Marshall JC, Namendys-Silva SA, et al. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014;2(5):380-386. doi:10. 1016/S2213-2600(14)70061-X.

[3] Jawad I, Lukšić I, Rafnsson SB. Assessing available information on the burden of sepsis:

- global estimates of incidence, prevalence and mortality. J Glob Health. 2012;2(1):010404. doi:10.7189/jogh.02.010404.
- [4] Evans L, Rhodes A, Alhazzani W, et al. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021;47(11):1181-1247. doi:10.1007/s00134-021-06506-y
- [5] Oh W, Takkavatakarn K, Kittrell H, Shawwa K, Gomez H, Sawant AS, Tandon P, Kumar G, Sterling M, Hofer I, Chan L, Oropello J, Kohli-Seth R, Charney AW, Kraft M, Kovatch P, Kellum JA, Nadkarni GN, Sakhuja A. Personalized Fluid Management in Patients with Sepsis and AKI: A Policy Tree Approach. medRxiv [Preprint]. 2025 Jan 23:2024.08.06.24311556. doi: 10.1101/2024.08.06.24311556. PMID: 39148835; PMCID: PMC11326317.
- [6] Morton Hamer MJ, Faught SK. Is Early Goal-Directed Therapy or Standard Therapy More Effective in Decreasing Mortality Among Patients With Sepsis? Ann Emerg Med. 2018 Jan;71(1):37-39. doi: 10.1016/j.annemergmed.2017.06.006. Epub 2017 Jul 14. PMID: 28712609.
- [7] Musikatavorn K, Plitawanon P, Lumlertgul S, et al. Randomized Controlled Trial of Ultrasound-guided Fluid Resuscitation of Sepsis-Induced Hypoperfusion and Septic Shock. West J Emerg Med. 2021;22(2):369-378. Published 2021 Feb 10. doi:10.5811/westjem.2020.11.48571
- [8] Verras C, Ventoulis I, Bezati S, Matsiras D, Parissis J, Polyzogopoulou E. Point of Care Ultrasonography for the Septic Patient in the Emergency Department: A Literature Review. J Clin Med. 2023; 12(3):1105. Published 2023 Jan 31. doi:10.3390/jcm12031105
- [9] Lee JY, Kim JY, Choi CH, Kim HS, Lee KC, Kwak HJ. The ability of stroke volume variation measured by a noninvasive cardiac output monitor to predict fluid responsiveness in mechanically ventilated children. Pediatr Cardiol. 2014 Feb;35(2):289-94. doi: 10.1007/s00246-013-0772-7. Epub 2013 Aug 21. PMID: 23963186.
- [10] Awadhare P, Patel R, McCallin T, Mainali K, Jackson K, Starke H, Bhalala U. Non-invasive Cardiac Output Monitoring and Assessment of Fluid Responsiveness in Children With Shock in the Emergency Department. Front Pediatr. 2022 Apr 7;10:857106. doi: 10.3389/fped.2022.857106. PMID: 35463892; PMCID: PMC9021702.
- [11] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. PMID: 24141714.
- [12] Nguyen HB, Rivers EP, Havstad S, Knoblich B, Ressler JA, Muzzin AM, Tomlanovich MC. Critical care in the emergency department: A physiologic assessment and outcome evaluation. Acad Emerg Med. 2000 Dec;7(12):1354-61. doi: 10.1111/j.1553-2712.2000.tb00492.x. PMID: 11099425.

- [13] Feissel M, Michard F, Faller JP, Teboul JL. The respiratory variation in inferior vena cava diameter as a guide to fluid therapy. Intensive Care Med. 2004 Sep;30(9):1834-7. doi: 10.1007/s00134-004-2233-5. Epub 2004 Mar 25. PMID: 15045170.
- [14] Mukherjee M, Rudski LG, Addetia K, Afilalo J, D'Alto M, Freed BH, Friend LB, Gargani L, Grapsa J, Hassoun PM, Hua L, Kim J, Mercurio V, Saggar R, Vonk-Noordegraaf A. Guidelines for the Echocardiographic Assessment of the Right Heart in Adults and Special Considerations in Pulmonary Hypertension: Recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2025 Mar;38(3):141-186. doi: 10.1016/j.echo.2025.01.006. Erratum in: J Am Soc Echocardiogr. 2025 Jul;38(7):641. doi: 10.1016/j.echo.2025.05.001. PMID: 40044341.
- [15] Rudski LG, Lai WW, Afilalo J, et al. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010;23(7):685-788. doi:10. 1016/j.echo.2010.05.010
- [16] Lichtenstein DA, Mezière GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol [published correction appears in Chest. 2013 Aug;144(2):721]. Chest. 2008; 134(1):117-125. doi:10.1378/chest.07-2800
- [17] Iwakura K, Onishi T. A practical guide to the lung ultrasound for the assessment of congestive heart failure. J Echocardiogr. 2021; 19(4):195-204. doi:10.1007/s12574-021-00528-7
- [18] Bentzer P, Griesdale DE, Boyd J, MacLean K, Sirounis D, Ayas NT. Will This Hemodynamically Unstable Patient Respond to a Bolus ofIntravenous Fluids? JAMA. 2016 Sep 27;316(12):1298-309. doi: 10.1001/jama.2016.12310. PMID: 27673307.
- [19] Monnet X, Marik P, Teboul JL. Passive leg raising for predicting fluid responsiveness: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1935-1947. doi: 10.1007/s00134-015-4134-1. Epub 2016 Jan 29. PMID: 26825952.
- [20] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID: 12065368.
- [21] Oord M, Olgers TJ, Doff-Holman M, Harms MP, Ligtenberg JJ, Ter Maaten JC. Ultrasound and NICOM in the assessment of fluid responsiveness in patients with mild sepsis in the emergency department: a pilot study. BMJ Open. 2017 Jan 27;7(1):e013465. doi: 10.1136/bmjopen-2016-013465. PMID: 28132006; PMCID: PMC5278240.
- [22] Chukwulebe SB, Gaieski DF, Bhardwaj A, Mulugeta-Gordon L, Shofer FS, Dean AJ. Early hemodynamic assessment using NICOM in patients at risk of developing Sepsis immediately after emergency department triage. Scand J Trauma Resusc Emerg Med.

- 2021;29(1):23. Published 2021 Jan 28. doi:10. 1186/s13049-021-00833-1
- [23] Zhu G, Zhang K, Fu Y, Hu Z. Accuracy assessment of noninvasive cardiac output monitoring in the hemodynamic monitoring in critically ill patients. Ann Palliat Med. 2020 Sep;9(5):3506-3512. doi: 10.21037/apm-20-1731. PMID: 33065801.
- [24] Min JJ, Lee JH, Hong KY, Choi SJ. Utility of stroke volume variation measured using non-invasive bioreactance as a predictor of fluid responsiveness in the prone position. J Clin Monit Comput. 2017 Apr;31(2):397-405. doi: 10.1007/s10877-016-9859-z. Epub 2016 Mar 10. PMID: 26964992.
- [25] Oord M, Olgers TJ, Doff-Holman M, Harms MP, Ligtenberg JJ, Ter Maaten JC. Ultrasound and NICOM in the assessment of fluid responsiveness in patients with mild sepsis in the emergency department: a pilot study. BMJ Open. 2017;7(1):e013465. Published 2017 Jan 27. doi:10. 1136/bmjopen-2016-013465
- [26] Cai XE, Ling WT, Cai XT, Yan MK, Zhang YJ, Xu JY. Effect of restrictive fluid resuscitation on severe acute kidney injury in septic shock: a systematic review and meta-analysis. BMJ Open. 2025 Feb 16; 15(2):e086367. doi: 10. 1136/bmjopen-2024-086367. PMID: 39956601; PMCID: PMC11831265.
- [27] Shahnoor H, Divi R, Addi Palle LR, Sharma A, Contractor B, Krupanagaram S, Batool S, Ali N. The Effects of Restrictive Fluid Resuscitation on the Clinical Outcomes in Patients with Sepsis or Septic Shock: A Meta-Analysis of Randomized-Controlled Trials. Cureus. 2023 Sep 20; 15(9):e45620. doi: 10.7759/cureus.45620. PMID: 37868575; PMCID: PMC10588294.
- [28] Toledo-Palacios HA, Pérez-Nieto OR, Reyes-Monge R, Rodríguez-Guevara I, Mark NM. Sepsis Resuscitation: Time to Embrace a Restrictive Fluid Strategy? J Am Coll Emerg Physicians Open. 2025 Jan 21;6(2):100040. doi: 10.1016/j.acepjo.2024.100040. PMID: 39895809; PMCID: PMC11780708.
- [29] Reynolds PM, Stefanos S, MacLaren R. Restrictive resuscitation in patients with sepsis and mortality: A systematic review and meta-analysis with trial sequential analysis. Pharmacotherapy. 2023 Feb;43(2):104-114. doi: 10.1002/phar.2764. Epub 2023 Jan 21. PMID: 36625778; PMCID: PMC10634281.
- [30] Devia Jaramillo G, Menendez Ramirez S. USER Protocol as a Guide to Resuscitation of the Patient with Septic Shock in the Emergency Department. Open Access Emerg Med. 2021; 13:33-43. Published 2021 Feb 12. doi:10.2147/OAEM.S289148
- [31] Verras C, Ventoulis I, Bezati S, Matsiras D, Parissis J, Polyzogopoulou E. Point of Care Ultrasonography for the Septic Patient in the Emergency Department: A Literature Review. J Clin Med. 2023; 12(3):1105. Published 2023 Jan 31. doi:10.3390/jcm12031105
- [32] Rice JA, Brewer J, Speaks T, Choi C, Lahsaei P, Romito BT. The POCUS Consult: How Point of Care Ultrasound Helps Guide Medical Decision Making. Int J Gen Med.

- 2021; 14:9789-9806. Published 2021 Dec 15. doi:10.2147/IJGM.S339476
- [33] Rice JA, Brewer J, Speaks T, Choi C, Lahsaei P, Romito BT. The POCUS Consult: How Point of Care Ultrasound Helps Guide Medical Decision Making. Int J Gen Med. 2021 Dec 15;14:9789-9806. doi: 10.2147/IJGM.S339476. PMID: 34938102; PMCID: PMC8685447.
- [34] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. PMID: 24171518.
- [35] Bateman RM, Sharpe MD, Jagger JE, 36th International Symposium on Intensive Care and Emergency Medicine: Brussels, Belgium. 15-18 March 2016. Crit Care. 2016 Apr 20;20(Suppl 2):94. doi: 10.1186/s13054-016-1208-6. Erratum in: Crit Care. 2016 Oct 24;20:347. doi: 10.1186/s13054-016-1358-6. PMID: 27885969; PMCID: PMC5493079.
- [36] Douglas IS, Alapat PM, Corl KA, Exline MC, Forni LG, Holder AL, Kaufman DA, Khan A, Levy MM, Martin GS, Sahatjian JA, Seeley E, SelfWH, Weingarten JA, Williams M, Hansell DM. Fluid Response Evaluation in Sepsis Hypotension and Shock: A Randomized Clinical Trial. Chest. 2020 Oct;158(4):1431-1445. doi: 10.1016/j.chest.2020.04.025. Epub 2020 Apr 27. PMID: 32353418; PMCID: PMC9490557.
- [37] Chaves RCF, Barbas CSV, Queiroz VNF, Serpa Neto A. Assessment of fluid responsiveness using pulse pressure variation, stroke volume variation, plethysmographic variability index, central venous pressure, and inferior vena cava variation in patients undergoing mechanical ventilation: a systematic review and meta-analysis. Crit Care. 2024 Aug 31;28(1):289. doi: 10.1186/s13054-024-05078-9. PMID: 39217370; PMCID: PMC11366151.
- [38] Awadhare P, Patel R, McCallin T, Mainali K, Jackson K, Starke H, Bhalala U. Non-invasive Cardiac Output Monitoring and Assessment of Fluid Responsiveness in Children With Shock in the Emergency Department. Front Pediatr. 2022 Apr 7;10:857106. doi: 10.3389/fped.2022.857106. PMID: 35463892; PMCID: PMC9021702.
- [39] Permpikul C, Leelayuthachai T. Non-invasive estimated continuous cardiac output (escCO) during severe sepsis and septic shock resuscitation. J Med Assoc Thai. 2014 Mar;97 Suppl 3:S184-8. PMID: 24772597.
- [40] Oord M, Olgers TJ, Doff-Holman M, Harms MP, Ligtenberg JJ, Ter Maaten JC. Ultrasound and NICOM in the assessment of fluid responsiveness in patients with mild sepsis in the emergency department: a pilot study. BMJ Open. 2017;7(1):e013465. Published 2017 Jan 27. doi:10. 1136/bmjopen-2016-013465